CLINICAL TRIAL: NCT04141358
Title: Using Ultrasound 2D Strain Speckle Tracking, 2D Shear Wave Elastography and Transonic Flowmeter as Diagnostic and Potential Predictor Tool for Arteriovenous Fistula Outcomes With End Stage Renal Failure.
Brief Title: Advanced Ultrasound Applications for Predicting AVF Outcomes
Acronym: AUAPAVFO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19HH5550
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: End Stage Renal Diseases; Renal Failure; Chronic Kidney Diseases
Keywords: Vascular Access; Endothelial Dysfunction; Vascular Stiffness; Arteriovenous Fistula
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — The leftover vessel specimens will be collected at the AVF surgery and placed immediately in a suitable biopsy container with formalin to prevent specimen drying. To study pre-existing diseases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with end-stage renal disease who will undergo arteriovenous fistula (AVF) surgery will be recruited and follow-up them up to 6 weeks or until the AVF become suitable for hemodialysis.
  Interventions: Diagnostic Test: Advanced ultrasound measurements

INTERVENTIONS:
Diagnostic Test: Advanced ultrasound measurements — Clinical interventions and procedures:
  * Consent at 0 week
  * Clinical data collection at 0 week
  * Strain for native artery at 0 week
  * Young's modulus for native artery at 0 week
  * Intimal medial thickness for native artery at 0 week
  * Ultrasound blood volume flow measurement at 0 week
  * Vessel diameter at 0 week
  * Blood pressure at 0 week
  * BMI at 0 week
  * Intra-operative blood volume flow measurement at AVF surgery time
  * Strain for native artery at 6 weeks
  * Young's modulus native artery at 6 weeks
  * Intimal medial thickness native artery arteries at 6 weeks
  * Ultrasound blood volume flow measurement at 6 weeks
  * Vessel diameter at 6 weeks
  * Blood pressure at 6 weeks
  * BMI at 6 weeks

SUMMARY:
Haemodialysis is a renal replacement therapy that can be introduced to patients with end-stage renal disease (ESRD) to help them maintain a good healthy life. The patient's blood is pumped through a dialysis machine to remove excess fluid, salt and waste, then it is pumped back into the patient's circulation system. In order to carry out haemodialysis, vascular access (VA) is required to connect the patient to the dialysis machine. Patients have only three options of vascular access: arteriovenous fistula (AVF), an anastomosis between a native vein and an artery; arteriovenous graft (AVG), a connection between a synthetic tube and native blood vessels; and (3) central line, a cuffed catheter placed in a large neck vein. Arteriovenous fistulas are the preferred method for VA because of their longevity and causing the least number of complications. Although there are a number of factors that may increase the probability of AVF failure rate such as age and gender of the patient, poor native vessel structure, medications and the level of surgical experience, 30-40% of new AVFs fail to mature for unknown reasons. For an AVF to become functionally mature postoperative, remodelling and dilation of the native artery and vein are essential to accommodate significantly increased blood flow. However, pre-existing diseases in patients with ESRD such as arterial stiffness and endothelial dysfunction may impair AVF and preclude dialysis. It has been asserted that the lack of AVF success is attributable to insufficient arterial dilation because of poor arterial wall elasticity.

The study aims to investigate the role of arterial stiffness and endothelial dysfunction in predicting AVF outcome using novel non-invasive ultrasound applications: 2D shear wave elastography and 2D strain speckle tracking will be employed to assess arterial stiffness, while an intraoperative flow-mediated dilation (FMD) technique will be used to evaluate endothelial dysfunction.

DETAILED DESCRIPTION:
This is an observational prospective pilot study of patients with end-stage renal disease (ESRD), who will be referred for AVF procedure.

Duration: 21 Months The research team will collect data from the patients after they have signed the informed consent form. Data collection will take place before, during and after arteriovenous fistula (AVF) surgery.

At 0 week, the patient will be interviewed to obtain clinical information. Also, blood pressure and body mass index will be checked and recorded. Next, pre-operative AVF assessment ultrasound measurements will be performed to assess flow, pulsatility and vessel diameter. Advanced ultrasound applications(2D strain speckle tracking and 2D Shear wave elastography) will be applied to assess arterial stiffness as additional measurement tools. These are quantitative measures of vessel stiffness. It takes less than five minutes to obtain these measurements from the imaged vessel.

During AVF surgery, the endothelial function will be assessed intraoperatively by testing the ability of the endothelium to dilate, flow mediation dilation (FMD). Leftover vessel specimens will be collected for histopathological analysis purpose.

At 6 week, post-AVF ultrasound assessment will be conducted to assess the maturation of AVF by measuring ultrasound parameters of blood flow, pulsatility and vessel diameter. Arterial stiffness parameters will be measured as well. Blood pressure and BMI will be assessed and recorded.

Study data will be entered into a study database which will consist of a password encrypted stored on a password-protected computer in the vascular lab at Hammersmith Hospital. Only the study researchers will know the study database password.

Data analysis will be performed after the enrolment of 20, 40 and 75 patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years age
* <90 years age
* End stage renal disease
* Glomerular filtration rate < 30 ml/min/1.73m2

Exclusion Criteria:

* <18 years age
* > 90 years age
* < 2cm vein diameter
* Not end-stage renal disease
* Pregnant patients will not be recruited in this study. Patients pregnancy status will be assessed on initial enrolment to exclude them from the study.
* Those unable to provide consent.
* Anyone who is taking part in any other research.
* Potential participants who might not adequately understand verbal explanations or written information given in English, or who have special communication needs will not be included

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients selected for this protocol must have the necessity to undergo surgery to receive an Arterio-Venos Fistula (AVF) for hemodialysis in either arm.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Patency of arteriovenous fistula according to ultrasound parameters | 6 Weeks
  Rate of blood volume flow >400 mL/min.
Arteriovenous fistula diameter | 6 Weeks
  Fistula considered to be patent if there is a minimum venous diameter of ≥ 5 mm.

SECONDARY OUTCOMES:
Number of arteriovenous fistula successful use for haemodialysis. | 10 weeks
  ≥ 3 uses on separate occasions post-arteriovenous fistula surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aslam, PhD, Study Director — Academic Supervisor
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kheda MF, Brenner LE, Patel MJ, Wynn JJ, White JJ, Prisant LM, Jones SA, Paulson WD. Influence of arterial elasticity and vessel dilatation on arteriovenous fistula maturation: a prospective cohort study. Nephrol Dial Transplant. 2010 Feb;25(2):525-31. doi: 10.1093/ndt/gfp462. Epub 2009 Sep 15. PMID 19755475
- [Background] McGrogan DG, Maxwell AP, Khawaja AZ, Inston NG. Current tools for prediction of arteriovenous fistula outcomes. Clin Kidney J. 2015 Jun;8(3):282-9. doi: 10.1093/ckj/sfv019. Epub 2015 Apr 2. PMID 26034589
- [Background] Owens CD, Wake N, Kim JM, Hentschel D, Conte MS, Schanzer A. Endothelial function predicts positive arterial-venous fistula remodeling in subjects with stage IV and V chronic kidney disease. J Vasc Access. 2010 Oct-Dec;11(4):329-34. doi: 10.5301/jva.2010.5833. PMID 21038305